CLINICAL TRIAL: NCT05539144
Title: A New Delineation Approach for Oral Cavity, Oropharynx, Larynx and Hypopharynx in Intensity-modulated Radiation Treatment for Head and Neck Cancer
Brief Title: A New Delineation Approach for Oral Cavity, Oropharynx, Larynx and Hypopharynx in IMRT for Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Provincial Hospital of Traditional Chinese Medicine (Other Government)
Responsible Party: Principal Investigator, Xueqi Wang, Principal Investigator, Hebei Provincial Hospital of Traditional Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HebeiProvincial
Record Dates: First submitted 2022-09-05; First posted 2022-09-14 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Head and Neck Cancer; Radiotherapy; Oropharynx Abnormality; Radiotherapy; Adverse Effect
Keywords: Oropharynx; Dosimetric parameters; Intensity-modulated radiation treatment（IMRT）; Head and Neck Cancer; Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "Oropharyngeal mucosa" as OARs (Experimental): "Oropharyngeal mucosa" was delineated as OARs and limiting its dose
  Interventions: Radiation: "Oropharyngeal mucosa"
- oropharynx as OARs (Experimental): Oropharynx was delineated as OARs and limiting its dose
  Interventions: Radiation: oropharynx
- Oropharynx and "oropharyngeal mucosa"as OARs (Experimental): Oropharynx and "oropharyngeal mucosa" was delineated as OARs and limiting its dose
  Interventions: Radiation: oropharynx and "oropharyngeal mucosa"

INTERVENTIONS:
Radiation: "Oropharyngeal mucosa" — "Oropharyngeal mucosa" was delineated as OARs and limiting its dose
  Arms: "Oropharyngeal mucosa" as OARs
Radiation: oropharynx — oropharynx was delineated as OARs and limiting its dose
  Arms: oropharynx as OARs
Radiation: oropharynx and "oropharyngeal mucosa" — oropharynx and "oropharyngeal mucosa"were delineated as OARs and limiting its dose
  Arms: Oropharynx and "oropharyngeal mucosa"as OARs

SUMMARY:
The investigators tries a new method to delineating the oral cavity, oropharynx, larynx and hypopharynx, and use the head-and-neck region to test whether the method can to create a good IMRT plan, and alleviate the oral radiation injury, reduce the incidence of adverse reactions.

DETAILED DESCRIPTION:
Purpose: To assess the dosimetric effect of new delineation approach for oral cavity, oropharynx, larynx and hypopharynx in intensity-modulated radiotherapy(IMRT) treatment planning for head and neck cancer.

Methods: Twenty head and neck cancer patients were treated by IMRT. Target volumes and several organs at risk were delineated with Corvus6．3 treatment planning system. An investigative IMRT plan was generated based on a standard treatment planning protocol, but used a new delineation approach for oral cavity, oropharynx, larynx and hypopharynx. Plans were exported to treatment planning system for quantitative analysis of dose volume parameters. Variables assessed included: maximum oral cavity, oropharynx, larynx and hypopharynx dose, equivalent uniform dose of the oral cavity, oropharynx, larynx and hypopharynx (EUD), mean oral cavity, oropharynx, larynx and hypopharynx dose, mean organs at risks (OARs) doses, and dose homogeneity inside the target volumes.

.

ELIGIBILITY:
Inclusion Criteria:

- patients with previously untreated of the head and neck cancer who received definitive IMRT at our institution

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Dose distribution | through study completion, an average of 1 year
  maximum oral cavity, oropharynx, larynx and hypopharynx dose, equivalent uniform dose of the oral cavity, oropharynx, larynx and hypopharynx (EUD), mean oral cavity, oropharynx, larynx and hypopharynx dose, mean organs at risks (OARs) doses, and dose homogeneity inside the target volumes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiotherapy, Hebei Province Hospital of Chinese Medicine, Shijiazhuang, Hebei, China